CLINICAL TRIAL: NCT04780464
Title: a 3 Arm Randomized Study on Health-related Quality of Life of Elderly Patients With Advanced Soft Tissue Sarcoma Undergoing Doxorubicin Alone Every Three Weeks or Doxorubicin Weekly or Cyclophosphamide Plus Predniso(lo)ne Treatment
Brief Title: A 3 Arm Randomized Study on Health-related QoL of Elderly Patients With Advanced Soft Tissue Sarcoma
Acronym: Tolerance
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Withdrawal grant provider
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1976-STBSG; 2021-000125-27 (EudraCT Number)
Record Dates: First submitted 2021-03-02; First posted 2021-03-03 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Advanced Soft-tissue Sarcoma
Keywords: Quality of Life; Elderly
MeSH Terms: interventions — Doxorubicin; Prednisolone; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard doxorubicin (Active Comparator)
  Interventions: Drug: Doxorubicin
- Metronomic doxorubicin (Experimental)
  Interventions: Drug: Doxorubicin
- Metronomic oral cyclophosphamide + prednisolone or prednisone (Experimental)
  Interventions: Drug: Cyclophosphamide Oral Product; Drug: Prednisolone; Drug: Prednisone

INTERVENTIONS:
Drug: Doxorubicin — 60 to 75 mg/m² intravenous, every 3 weeks for max 6 cycles until PD
  Other Names: Adriamycin;
  Arms: Standard doxorubicin
Drug: Doxorubicin — 12 mg/m2 intravenous weekly for a maximum of 450 mg/m2 until PD
  Other Names: Adriamycin;
  Arms: Metronomic doxorubicin
Drug: Cyclophosphamide Oral Product — 100 mg BD on day 1 to day 7 of each 14 day cycle until PD
  Arms: Metronomic oral cyclophosphamide + prednisolone or prednisone
Drug: Prednisolone — 10-20 mg on day 1 to day 7 of each 14 day cycle until PD
  Arms: Metronomic oral cyclophosphamide + prednisolone or prednisone
Drug: Prednisone — 10-20 mg on day 1 to day 7 of each 14 day cycle until PD for those Countries where Prednisolone in tablets is not available
  Arms: Metronomic oral cyclophosphamide + prednisolone or prednisone

SUMMARY:
This is a multi-centre, open label, randomized phase 3 selection study (1:2:2 randomization).

After confirmation of the eligibility criteria, 185 patients will be randomized 1:2:2 to either the control arm (doxorubicin 60-75 mg/m² IV every 3 weeks) or experimental arm 1 (doxorubicin 12 mg/m2 IV every week) or experimental arm 2 (cyclophosphamide 100 mg orally BD plus prednisolone 10-20 mg orally on day 1 to day 7 of each 14 day cycle).

HRQoL assessment will be performed every 3 weeks during the first 12 weeks and every 12 weeks thereafter until month 12 after start of treatment.

Disease evaluation will be performed every 12 weeks until progression. The primary endpoint of the study is difference among the study arms in physical and role functioning at 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven advanced unresectable or metastatic soft tissue sarcoma
* Representative formalin fixed, paraffin embedded tumor blocks or a minimum of 10 unstained tissue slides, either from the primary tumor or a metastatic lesion, must be available for histological central review. Histological central review is not required before treatment start but it is mandatory to send at least 10 unstained tumor slides (blocks optional) at time of study entry. Local histopathological diagnosis will be accepted for entry into this trial.
* Age ≥ 65 years of age (patients between 65 and 69 years old are eligible if G8 score ≤ 14; patients ≥ 70 years old are eligible independent of G8 score)
* WHO performance status 0 - 2
* Life expectancy based on other significant morbidity of ≥ 6 months
* Presence of measurable disease (according to RECIST 1.1), as confirmed by imaging within the 28 days prior to randomization. CT with IV contrast is the preferred imaging modality. In case of any contra-indications (medical or regulatory), it is allowed to perform a non-contrast CT + MRI.
* Progressive disease at entry based on RECIST 1.1
* Patients amenable to receive doxorubicin according to investigator's assessment
* Adequate haematological and organ function assessed prior to randomization:
* Haematological function:

  * haemoglobin ≥ 9.0 g/dL or 5.6 mmol/L
  * absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * platelet count ≥ 100 x 109/L
  * Coagulation: partial thromboplastin time (PTT) ≤ 1.0 times upper limit of normal (1.0 x ULN) of institutional limits and prothrombin time (PT) ≤ 1.0 x ULN of institutional limits
* Renal function: estimated glomerular filtration rate (eGFR) > 50 ml/min/m2 (calculated by the MDRD formula in appendix E); no proteinuria ≥ grade 2 (CTCAE version 5.0);
* Hepatic function: bilirubin ≤ 1.0 x ULN of institutional limits, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤1.5 x ULN.

If isolated elevated bilirubin <2 x ULN and Gilberts syndrome suspected, suggest repeating bloods after food. If bilirubin improves to meet the criteria above this is acceptable. More severe persistent hepatic impairment of whatever cause would exclude the patient from treatment till resolved.

* Cardiac function: clinically normal function based on the institutional lower limit of normal for left ventricular ejection fraction (LVEF) as assessed either by multi-gated acquisition scan (MUGA) or cardiac ultrasound and 12 lead electrocardiogram (ECG) without clinically relevant abnormalities. Measurement should include investigator assessment of a potential participant's risk for heart failure with a validated clinical classification system, i.e. the New York Heart Association Functional Classification. Only patients with NYHA class 1 and 2 according to appendix D are eligible.
* Completion of EORTC QLQ-C30 and EORTC QLQ-ELD14 at baseline.
* Assessment of G8 geriatric screening tool
* Assessment of Katz Index of Independence in Activities of Daily Living (ADL)
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:
* With female partners of childbearing potential, men must remain abstinent or use a condom during the treatment period and for a period of 6 months after the last dose of doxorubicin-based chemotherapy and for a period of 12 months after the last dose of cyclophosphamide-based chemotherapy. Men must refrain from donating sperm during this same period. Contraception should be considered for the female partners of childbearing potential as well.
* With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for a period of 6 months after the last dose of doxorubicin-based chemotherapy and for a period of 12 months after the last dose of cyclophosphamide-based chemotherapy to avoid exposing the embryo.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations including commitment to completing questionnaires during the course of the study.

Exclusion Criteria:

* Symptomatic or known brain metastasis
* Any prior treatment with anthracyclines
* Any prior systemic treatment for metastatic STS
* Inability to swallow and/ or retain oral tablets
* Rare hereditary galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Hypersensitivity to doxorubicin, cyclophosphamide, prednisolone or to any of their metabolites or to any of their excipients
* Uncontrolled severe illness, including but not limited to:
* Congestive heart failure
* Angina pectoris
* Acute inflammatory heart disease
* Myocardial infarction within 1 year before randomization
* Arterial hypertension defined as blood pressure ≥ 150/100 mm Hg despite optimal medical therapy
* Uncontrolled cardiac arrhythmia
* Increased haemorragic tendency
* Uncontrolled diabetes
* Bone marrow aplasia
* Psychosis
* Active or uncontrolled infections among which those requiring systemic antibiotics or antimicrobial therapy.
* Inflammation of the urinary bladder (interstitial cystitis) and/or obstructions of the urine flow.
* Vaccination with live vaccines within 30 days prior to study entry
* Patients with a prior or concurrent malignancy whose natural history or treatment has the potential to interfere with the safety or efficacy assessment of the investigational regimen are not eligible for this trial.
* Known contraindication to imaging tracer or contrast medium and contraindication to MRI
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and its active requirements (including completion of questionnaires) and follow-up schedule; those conditions should be discussed with the patient before randomization in the trial

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-11-11 (Actual)

PRIMARY OUTCOMES:
Health-related Quality of Life | 4 years after first patient in
  Difference in physical and role functioning at 12 weeks

SECONDARY OUTCOMES:
Tumour response | 5.5 years after first patient in
  tumor response according to RECIST criteria (version 1.1)
Progression-free-survival | 5.5 years after first patient in
  Progression-free-survival from the date of randomization to the date of first progression or death, whatever comes first
Overall survival | 5.5 years after first patient in
  Overall survival from the date of randomization to the date of death, whatever the cause

CONTACTS AND LOCATIONS:
Overall Officials: Winette van der Graaf, Study Chair — Nationaal Kanker Instituut, Amsterdam, NL
Locations (2):
- Bank Of Cyprus Oncology Centre, Nicosia, Cyprus
- King Hussein Cancer Center, Amman, Jordan